CLINICAL TRIAL: NCT03081325
Title: A Preliminary Study About Unexplained Recurrent Miscarriage and Repeated Implantation Failure Patients Treated With Low-dose Lymphocyte Immunotherapy
Acronym: immunotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Principal Investigator, Nanjing University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL2015007
Record Dates: First submitted 2017-03-08; First posted 2017-03-16 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Unexplained Recurrent Miscarriage and Recurrent Implantation Failure
Keywords: uRM; RIF; Th1; Th2; Treg; lymphocyte immunotherapy

ARMS (1):
- lymphocyte immunotherapy on uRM and RIF (Experimental): Donor (husband or third party) lymphocytes were prepared by Ficoll-Paque centrifugation; the cells were washed with sterile saline and resuspended in 1 ml at a concentration of 20-40 × 106 cells/ml. The cells were given to the female partner by 4-6 intradermal injected. In this study, the lymphocyte immunization therapies were performed every 3 weeks for 3 times. After that we test Th1/Th2/Treg, if they become normal, the patients can prepare for pregnancy.
  Interventions: Procedure: low-dose lymphocyte immunotherapy

INTERVENTIONS:
Procedure: low-dose lymphocyte immunotherapy — Peripheral venous blood (PBMCs) was drawn from the husbands of uRM and RIF patients and then the PBMCs were resuspended and administered intradermally to uRM and RIF patients 3 times at 3-week intervals. Once conceived, the uRM and RIF patients undergo 2 rounds of treatment at 8-week intervals.

SUMMARY:
Recurrent miscarriage(RM) and recurrent implantation failure (RIF) are clinical challenge for clinicians and patients who are desperate for a healthy child.The specific etiology contains chromosomal abnormalities, reproductive anatomical abnormalities, endocrine disorders, reproductive system infections, autoimmune and environmental factors. However there are still 50% to 60% RM and RIF which don't have a clear cause,mainly associated with alloimmune factors.Among various treatments,lymphocytes active immunotherapy is the most common treatment method, and its clinical efficacy is widely recognized although its action mechanism is not clear so far.

DETAILED DESCRIPTION:
The main mechanism of active immunotherapy includes upregulating Th2-type cytokines, downregulating Th1-type cytokines, making Th1 / Th2 shift to Th2, inducing maternal serum IL-6 and sIL6R, PIBF, EGF; inducing the expression of Fas / Fasl on lymphocyte surface; increasing the proportion of CD8 + cells, Th2-type cells and CD + CD25 + Treg cells, decreasing the activity of CD56 + CD16 + NK cell and so on.The purpose of this study is to observe the treatment effects of active immunotherapy on uRM and RIF patients. What's more,we will used flow cytometry, and quantitative real-time PCR (qPCR) methods to characterize Th1、Th2 and Treg cell populations after immunotherapy,ecpecting to find out the exact molecule mechanism of immunotherapy with paternal or third party lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy except for their history of recurrent abortions and were negative for blocking antibodies
* Willing to receive follow up

Exclusion Criteria:

* Patients with genetic impairment
* Patients with Mullerian anomaly
* Patients with hormonal deficiency
* Patients with metabolic disorder
* Patients with infectious disease
* Patients with autoimmune abnormalities

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
T cell proportion | 1 year
  We use flow cytometry to detecte peripheral blood Th1、Th2 and Treg cells of uRM and RIF patients before and after low-dose lymphocyte immunotherapy to see if the immunotherapy have treatment effect on Th1/Th2/Treg paradigm disorder
Abortion rate | 1 year
  We undergo follow-up of all the uRM patients to see the abortion rate (miscarriage was confirmed by ultrasound before the 20th week of gestation) after lymphocyte immunotherapy
IVF outcomes | 1 year
  We observed the the implantation rate, clinical pregnancy rate, and ongoing pregnancy rate of RIF patients after low-dose lymphocyte immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu M, Zhen X, Song H, Chen J, Sun X, Li X, Zhou J, Yan G, Ding L, Sun H. Low-dose lymphocyte immunotherapy rebalances the peripheral blood Th1/Th2/Treg paradigm in patients with unexplained recurrent miscarriage. Reprod Biol Endocrinol. 2017 Dec 16;15(1):95. doi: 10.1186/s12958-017-0315-9. PMID 29246150